CLINICAL TRIAL: NCT02973230
Title: Serum Vascular Endothelial Growth Factor (VEGF) As a Marker for Tubal Pregnancy
Brief Title: Serum VEGF as a Tubal Pregnancy Marker
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Fábio Roberto Cabar, MD; MSc, PhD, University of Sao Paulo General Hospital
Other Study IDs: fcabarVEGF1
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy, Ectopic
Keywords: Pregnancy, Ectopic; Vascular Endothelial Growth Factor A; Pregnancy, Tubal
MeSH Terms: conditions — Pregnancy, Ectopic; Pregnancy, Tubal

INTERVENTIONS:
Other: Dosage of VEGF serum concentration — Blood samples were collected by peripheral venous puncture before treatment; a total 15 mL of blood was withdrawn (2 mL for β-hCG, 3mL for progesterone, 10 mL for VEGF determinations). Blood samples for VEGF were collected in siliconized tubes and were allowed to coagulate at room temperature for 2-6 hours.

SUMMARY:
The aim of the present study was (i) to evaluate whether a single measurement of VEGF would allow us to distinguish between intrauterine pregnancy (normal and abnormal) and EP and (ii) to correlate the levels of VEGF with serum levels of progesterone and β-hCG in each subgroup.

Ninety patients were selected from a population of women presenting to the Hospital das Clínicas of the University of São Paulo Medical School from October 2006 until September 2007 and were divided in three subgroups: (i) abnormal (arrested) intrauterine pregnancy (defined as a gestational sac greater than 16 mm of mean diameter without fetal tissue or a embryo greater than 5 mm without embryo cardiac activity); (ii) tubal pregnancy (no evidence of intrauterine pregnancy, presence of a adnexal mass, suboptimal rise of serum hCG levels in 48 hours); all tubal pregnancies were surgically treated and were histologically confirmed, they did not receive any methotrexate treatment before operation; (iii) normal intrauterine pregnancy (intrauterine gestational sac, embryo vitality confirmed).

Blood samples were collected by peripheral venous puncture before treatment; a total 15 mL of blood was withdrawn (2 mL for β-hCG, 3mL for progesterone, 10 mL for VEGF determinations). Blood samples for VEGF were collected in siliconized tubes and were allowed to coagulate at room temperature for 2-6 hours.

ELIGIBILITY:
Inclusion Criteria were:

* women that had a positive hCG test and presented with either abdominal pain or vaginal bleeding; all pregnancies were singletons, spontaneously conceived, with accurate assessments of their gestational age (42 - 56 days from the first day of the last menstrual period). A detailed informed consent was obtained from each patient before the inclusion.

Exclusion Criteria was:

* non-ampullar tubal pregnancy (surgically confirmed).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
VEGF serum concentration | One year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo - School of Medicine - General Hospital, São Paulo, São Paulo, Brazil